CLINICAL TRIAL: NCT00978159
Title: Esomeprazole or Famotidine in the Management of Aspirin Related Non-ulcer Dyspepsia - a Double Blind Randomized Control Study
Brief Title: Esomeprazole or Famotidine in the Management of Aspirin Related Non-Ulcer Dyspepsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruttonjee Hospital (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Fook-Hong Ng, CON, Ruttonjee Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKEC 2009-058
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Aspirin; Dyspepsia
Keywords: esomeprazole; famotidine; aspirin; dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Esomeprazole; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esomeprazole (Active Comparator): esomeprazole 20 mg
  Interventions: Drug: esomeprazole
- Famotidine (Active Comparator): famotidine 40 mg
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: esomeprazole — esomeprazole 20 mg po for 4 weeks
  Arms: esomeprazole
Drug: Famotidine — Famotidine 40 mg po for 4 weeks
  Arms: Famotidine

SUMMARY:
Aspirin can prevent ischemic vascular disease but is commonly complicated by dyspepsia in 30% of patients. Patients, who have aspirin related dyspepsia, commonly underwent upper endoscopy to exclude peptic ulcer disease or gastric cancers. For those without significant lesions in the stomach and duodenum (non-ulcer dyspepsia), the best approach in the management is unclear. The objective of this study is to compare the efficacy of esomeprazole and famotidine in the control of dyspeptic symptom. After giving consent, patients will be randomised to receive either esomeprazole 20 mg daily or famotidine 40 mg daily in a double blinded manner. The patient will be followed-up at the 2nd and 4th week. The study will be completed at the 4th week. The primary analysis will be the efficacy in the control of dyspepsia symptom between the two groups.

DETAILED DESCRIPTION:
The objective of this double blinded randomized controlled study is to compare the efficacy of esomeprazole with famotidine in the control of dyspepsia in patients with aspirin related nonulcer dyspepsia NUD.

Method

The study shall be applied for approval from the Ethic Committee of Hong Kong West and East Cluster and shall be registered to the Clinical Trial Governance before the recruitment of the first patient.

Measuring instruments & Definitions

Hong Kong Dyspepsia Index (HKDI)

The presence or absence of dyspepsia was measured by the validated Hong Kong index of dyspepsia . This questionnaire could be used in epidemiological studies assessing the frequency and severity of dyspepsia in patient populations and also in interventional studies in functional dyspepsia.This index consisted of 12 questions on the severity of gastrointestinal symptoms, graded according to a five-point Likert scale (1- 5, from asymptomatic to very severe symptoms). A cut-off score of equal to or greater than 16 was determined to discriminate between controls and dyspeptic patients.

Global Dyspepsia Score

The global severity of dyspepsia will be measured by the Global Dyspepsia Score, which was a four-point scale in which a score of 0 indicated no pain or discomfort, a score of 1 mild pain or discomfort, a score of 2 moderate (annoying but not interfering with the daily routine) pain or discomfort, and a score of 3 severe (markedly interfering with the daily routine) pain or discomfort over the last 7 days . This scale is reliable, valid, and responsive and provides global assessment of symptoms in the western population . Significant dyspepsia was defined when Global Dyspepsia Score was more than or equal to 2 moderate.

Definition of significant endoscopic finding

Significant finding was defined as the presence of reflux esophagitis, Barrett's esophagus, gastric or duodenal ulceration, duodenal or esophageal erosions, or cancer and those with more than five gastric erosions on upper endoscopy. (Tally N, NEJM 1999)

ELIGIBILITY:
Inclusion Criteria:

* at least moderate pain or discomfort (or both) centered in the upper abdomen as their predominant symptoms for 7 days before randomization; taking low dose aspirin (80-300 mg daily),and insignificant upper endoscopic finding. At least moderate pain or discomfort is defined if the HKDI was more than or equal to 16.
* H. Pylori: In patients with have successful eradication of H. pylori and had dyspepsia with HKDI >=16 at the 6th week after eradication therapy can be recruited.In patients without H. pylori infection, they can be recruited immediately.

Exclusion Criteria:

* non-Chinese speaking
* significant endoscopic finding
* typical biliary colic
* predominant heartburn or symptoms of the irritable bowel syndrome
* a history of peptic ulcer or gastroesophageal reflux
* unintentional weight loss previous gastric or duodenal surgery
* thrombocytopenia
* renal failure with estimated creatinine clearance less than 10 ml/min
* active cancer
* known allergic to aspirin, famotidine or esomeprazole
* pregnancy, lactation, child-bearing potential in the absence of contraception
* planned co-prescription of nonsteroidal anti-inflammatory drugs
* corticosteroid, clopidogrel or anticoagulant
* anxiety neurosis, depression, psychosomatic disorder
* investigation for dyspepsia with endoscopy or barium series before aspirin therapy or disorders that might modify the absorption of study drugs
* ongoing treatment with a histamine H2-receptor antagonist, a prostaglandin, or a prokinetic drug during the 7 days before enrollment was not permitted, nor was treatment with a proton-pump inhibitor, or bismuth in the 30 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Treatment success : The HKDI is less than 16. Treatment was considered to have failed if a patient had taken medication for dyspepsia (other than antacids) during the study period | 4 weeks

SECONDARY OUTCOMES:
Treatment success: no significant dyspepsia defined by the Global Dyspepsia Score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: FH Ng, MD, Principal Investigator — Ruttonjee Hospital
Locations (2):
- China (2):
  - Queen Mary Hospital, Pokfulam, Hong Kong
  - Ruttonjee Hospital, Hong Kong